CLINICAL TRIAL: NCT02981212
Title: Multi-center, Randomized, Open Label, Comparative, Phase IV Study to Evaluate the Efficacy and Safety of a Combination of Mycophenolate Mofetil and Corticosteroid for 48 Weeks in Advanced IgA Nephropathy
Brief Title: Efficacy and Safety of a Combination of Mycophenolate Mofetil and Corticosteroid in Advanced IgA Nephropathy
Acronym: AIGA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Collaborators: Chong Kun Dang Pharmaceutical Corp. (Industry); Kyung Hee University Hospital at Gangdong (Other); Kyungpook National University Hospital (Other); Pusan National University Yangsan Hospital (Other); Inje University (Other); Seoul St. Mary's Hospital (Other); Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Beom Seok Kim, Professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 062IGA15-1D
Record Dates: First submitted 2016-11-24; First posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-11

CONDITIONS: IgA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Mycophenolic Acid; Angiotensin-Converting Enzyme Inhibitors; Conservative Treatment; Adrenal Cortex Hormones; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mycophenolate Mofetil (Experimental): MYREPT® capsule(CKDpharm, KOREA) and corticosteroid
  Interventions: Drug: Mycophenolate Mofetil; Drug: Corticosteroid
- Conservative treatment (Active Comparator): maintain conservative treatment (ACE inhibitor or ARB)
  Interventions: Drug: ACE inhibitor; Drug: ARB

INTERVENTIONS:
Drug: Mycophenolate Mofetil — less than 80 kg: 1,500 mg / day , 80 kg or more: 2,000 mg / day divided twice a day and administered orally
  Other Names: MYREPT®
  Arms: Mycophenolate Mofetil
Drug: ACE inhibitor — maintain conservative treatment (using ACE inhibitor or ARB for blood pressure regulation and proteinuria suppression treatment) just as before randomization
  Other Names: conservative treatment
  Arms: Conservative treatment
Drug: Corticosteroid — combination with Mycophenolate Mofetil
  Other Names: prednisolone; methyprednisolone
  Arms: Mycophenolate Mofetil
Drug: ARB — maintain conservative treatment (using ACE inhibitor or ARB for blood pressure regulation and proteinuria suppression treatment) just as before randomization
  Other Names: conservative treatment
  Arms: Conservative treatment

SUMMARY:
The purpose of this clinical study is to evaluate the efficacy and safety of that test group was administered with Mycophenolate Mofetil in combination with corticosteroid in patients with advanced IgA nephropathy. The control group will be observed for up to 48 weeks without administration of Mycophenolate Mofetil.

DETAILED DESCRIPTION:
The subject who signed the written agreement to participate in the clinical trial evaluates the conformity and then 1: 1 randomly allocated.

The study group were taken 48 weeks with MYREPT ® capsules in combination with corticosteroids and the control group were asked to preserve the conservative treatment regimen prior to the clinical trial registration Maintenance.

The subject who started taking the study medicine will carry out the examination and procedure if it has to be carried out for the visit via outpatient clinic at 4 weeks, 12 weeks, 24 weeks, 36 weeks, 48 weeks.

ELIGIBILITY:
Inclusion Criteria

1. Patient aged 19 to 65 years old
2. Diagnosed with IgA nephropathy
3. Confirmed with Proteinuria more than 1.0 g / day at least twice within 6 months from the time of screening
4. If eGFR (by MDRD) is <50 mL / min / 1.73 m^2, ≥ 15 mL / min / 1.73 m^2
5. ACE inhibitor or ARB for at least 3 months
6. Willing and able to provide written informed consent.

Exclusion Criteria:

1. If eGFR (by MDRD) is <15 mL / min / 1.73 m^2
2. Blood pressure is SBP> 160 mmHg or DBP> 100 mmHg
3. Systemic infection or have been diagnosed with cancer within the last 5 years (excluding treatment squamous cell or basal cell carcinoma skin cancer)
4. serious digestive disorder
5. WBC <3000 / mm^3
6. Acute (within 4 weeks) or chronic(need to treatments) allergic/hypersensitivity reaction in the history of Investigational drugs
7. Administration of other Investigational drugs within 28days before screening period
8. Administration of Investigator drug or other immunosuppressants within 84days before screening period
9. Women in pregnant or breast-feeding or don't using adequate contraception.
10. Patient has conversation impairment because alcohol or drugs addiction history within 6months or mental illness, etc.
11. In investigator's judgment

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-08 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Remission rate (complete / partial) | up to 48 weeks

SECONDARY OUTCOMES:
Remission rate (complete / partial) | at 12 weeks, at 24 weeks, at 36 weeks
eGFR(estimated glomerular filtration rate) by MDRD(modification of diet in renal disease) | at 24 weeks, at 36 weeks, at 48 weeks
The incidence of renal replacement therapy | up to 48 weeks
  renal replacement therapy; dialysis, new transplant
The average time to occurrence of renal replacement therapy | up to 48 weeks
  renal replacement therapy; dialysis, new transplant

CONTACTS AND LOCATIONS:
Overall Officials: BEOMSUK KIM, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No